CLINICAL TRIAL: NCT01760590
Title: The Effects of Thoracic Spine Manipulation and Mobilization in Individuals With Nontraumatic Cervical Pain
Brief Title: The Effects of Thoracic Spine Manipulation in Individuals With Non-traumatic Cervical Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keystone Rehabilitation Systems (Other)
Responsible Party: Principal Investigator, Joseph Brence, Co-Investigator, Keystone Rehabilitation Systems
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KRS2
Record Dates: First submitted 2012-12-22; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Neck Pain; Cervical Pain
Keywords: neck pain; cervical pain; pain pressure thresholds; pain catastrophizing
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations; Heimlich Maneuver

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual Manipulation (Experimental): Patients will be randomized to receive a thrust manipulation
  Interventions: Procedure: Manual Manipulation
- Manual Mobilization (Experimental): Patients will be randomized to receive mobilization
  Interventions: Procedure: Mobilization

INTERVENTIONS:
Procedure: Manual Manipulation — A grade 5 thrust to the thoracic spine
  Other Names: Thrust
  Arms: Manual Manipulation
Procedure: Mobilization — A grade 1-4 mobilization directed at thoracic spine
  Other Names: Springing
  Arms: Manual Mobilization

SUMMARY:
The purpose of this research is to compare the effects of two commonly used, safe, thoracic spine grade 1-4 and grade 5 mobilization to the thoracic spine on cervical spine pain in individuals with nontraumatic cervical pain. The immediate effects of thoracic spine mobilization have been shown to facilitate greater range of motion increases in the cervical spine and greater pain decreases within a treatment session and on follow-up visits. There is no research utilizing pain threshold perception as an objective outcome of these treatments. Only one study compared the two treatment techniques and concluded that future research should be completed which includes manual therapy for the thoracic spine. (Cleland 2007)

DETAILED DESCRIPTION:
The purpose of this research is to compare the effects of two commonly used, safe, thoracic spine grade 1-4 and grade 5 mobilization to the thoracic spine on cervical spine pain in individuals with nontraumatic cervical pain. The immediate effects of thoracic spine mobilization have been shown to facilitate greater range of motion increases in the cervical spine and greater pain decreases within a treatment session and on follow-up visits. There is no research utilizing pain threshold perception as an objective outcome of these treatments. Only one study compared the two treatment techniques and concluded that future research should be completed which includes manual therapy for the thoracic spine. (Cleland 2007)

The subjects will be patients at clinics owned by Physiotherapy Associates, Fit Physical Therapy, and Allegheny and Chesapeake PT who seek physical therapy services for nontraumatic neck pain. Participation will be entirely voluntary.

Patients will be offered a chance to participate in the research project on their initial visit for Physical Therapy.

If the PT identifies an appropriate patient they will ask if they are interested in being a research subject. The Physical Therapist recruiting subjects all have completed their Doctor of Physical Therapy Degree and have advanced training in manual Physical Therapy. The techniques employed are considered standard practice and are defined as entry level skills by the Commission of Accredidation of Physical Therapy Programs. These techniques are typically taught in DPT degree programs.

If the patient is interested, a description of the study will be provided. A consent form will be given to all participants.

Research Procedures:

1. Patients who present to one of three Physical Therapy clinics, under the direction of three advanced clinicians, will be assessed for their potential participation in this research. The treating clinician will recruit appropriate subjects based on includion and exclusion criteria and their PT diagnosis. Those that meet the inclusion and exclusion criteria will be given the consent form to determine if they wish to participate. Each researcher will have formal training in these techniques. Two of the clinicians have received their Orthopedic Clinical Specialists certification under the examination prcess outlined by the American Physical Therapy association. A third researcher has obtained his fellowship designation from the American Academy of Orthopedic Manual Physical Therapy. This skill is deemed entry level by the the Accredidation Board of the American Physical Therapy Educators. All Therapists will undergo a prestudy hands on education program to ensure the use of similar techniques.
2. If after reading the consent form they agree to participate, they will be given one additional form, the Pain Catastrophizing scale, and asked to complete it. The scale, NDI, cervical ROM, age, and birthdate will be recorded on a sheet contained in the patient's clinical chart.
3. The PT evaluation will then be completed.
4. They will then be randomized into one of two groups based on a roll of a die:

   Group One: Mobilization Group: this group will receive grade 1,2,3,or 4 mobilization in prone based on the PT's clinical judgement.

   The treatment parameters will be recorded.

   Group Two: Grade 5 mobilization group: this group wil receive a grade 5 mobilization.
5. Additional treatment including patient eduation, modalities, and exercise will be completed as the PT deems appropriate,
6. The second visit will be scheduled within 24 to 48 hours.
7. The patient will complete the same forms as were completed during the initial evaluation (NDI, PCS) and return them so that the results may berecorded on the record sheet identified only with date of birth.
8. The treatment will be repeated including the manual technique and other treatment deemed appropriate by the PT. Additional treatment between the second and last visits will be under the sole discretion on the treating PT.
9. On the discharge visit, the patient will receive the same forms, and be asked how much, in terms of %, they feel they have improved. This information will be recorded on the deidentified sheet.

Home exercise programs and patient educaiton will be issued as appropriate.

A bubble goniometer will be used for range of motion assessment. This is a standard plastic device used in PT practice. A Wagner FDX digital force gauge algometer will measure pain pressure thresholds.

Where survey instruments are involved, a copy of the instrument and, for surveys not created for this project, assurance that the principal investigator has proper approval to use them.

The Neck Disability Index or NDI will be used. It is the professional standard for outcomes measures for people with neck pain.

It has been shown to be valid and reliable.

The Pain Castrophizing Scale will be used. It is a valid and reliable measure of a patient's perception of pain and is commonly used.

The data will be collected by the treating Physical Therapist who has access to the patient record for treatment purposes.

The data will not be used for purposes other that patient care and research purposes.

Patient's data measures will be collected on a de-identified sheet marked with the patients birthday. The will be kept in a locked area in the clinic. The lead investigator will have access to the data when the study is completed and transfer it to a locked file cabinet in his office for data assessment.

Following treatment the patient may have mild soreness over the area which was treated. This typically diminishes in 24 hours. the patient will be informed of this potential soreness. The use of heat and /or ice, exercise, and patient education provided by the Therapist concerning activities and posture will also lessen the soreness.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients with non-traumatic Neck Pain
* Between ages 18 - 60

EXCLUSION CRITERIA:

Red flags such as:

* leg weakness
* night pain
* history of cancer
* upper motor neuron signs
* infection
* tumors
* osteoporosis
* fracture
* history of whiplash within 6 weeks
* cervical stenosis
* CNS involvement
* signs consistent with nerve root compression
* previous surgery
* pending legal action

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Pain | Baseline, change from baseline to week 1 and change from baseline to week 4 (discharge as per PTs discretion but typically 4 weeks)
  Verbal Descriptor on a scale from 0-10
Neck Disability | Baseline, change from baseline to week 1 and change from baseline to week 4 (discharge as per PTs discretion but typically 4 weeks)
  Neck Disability Index
Pain Pressure Thresholds | Baseline, change from baseline to week 1 and change from baseline to week 4 (discharge as per PTs discretion but typically 4 weeks)
  Using Wagner FDX Algometer

SECONDARY OUTCOMES:
Pain Catastrophizing | Baseline, change from baseline to week 1 and change from baseline to week 4 (discharge as per PTs discretion but typically 4 weeks)
  Pain Catastrophizing Scale
Global Rating of Change | Baseline will be assessed at Week 1 and change from this measurement taken at Week 4
  % of perceived change following intervention
ROM | Baseline, change from baseline to week 1 and change from baseline to week 4 (discharge as per PTs discretion but typically 4 weeks)
  Bubble goniometry of cervical motion
Clinical Equipoise | Baseline
  This will measure examiners C.E

CONTACTS AND LOCATIONS:
Overall Officials: Steve Karas, DSc, Study Director — Chatham University; Joseph B Brence, DPT, Principal Investigator — Keystone Rehabilitation Systems
Locations (2):
- United States (2):
  - Keystone Rehabilitation Systems, Bridgeville, Pennsylvania
  - Allegheny Chesapeake Physical Therapy, Pittsburgh, Pennsylvania